CLINICAL TRIAL: NCT03830190
Title: Cost-Effectiveness of Specialized Nursing Interventions for Patients With Parkinson's Disease
Brief Title: Cost-effectiveness of Nursing Interventions for Patients With PD
Acronym: NICE-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NICE-PD
Record Dates: First submitted 2018-12-20; First posted 2019-02-05 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2020-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Parkinson's disease nurse specialist; Nursing; Quality of life; Cost-effectiveness; Multidisciplinary care
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with 2 study arms: the intervention group and the control group. Participants are allocated to each arm in a 1:1 ratio.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the type of intervention (Parkinson's disease nurse specialist care), the participant and care provider cannot be masked. The investigator and outcome assessor (conducting the questionnaires) will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Parkinson's disease nurse specialist care
  Interventions: Other: Parkinson's disease nurse specialist care
- Control group (No Intervention): No intervention

INTERVENTIONS:
Other: Parkinson's disease nurse specialist care — Specialized nursing care provided by a Parkinson's disease nurse specialist
  Other Names: PDNS care
  Arms: Intervention group

SUMMARY:
Background: Current guidelines recommend that every person with Parkinson's disease (PD) should have access to Parkinson's Disease Nurse Specialist (PDNS) care. Thus, hospitals increasingly offer PDNS care to their patients with PD. However, there is currently little scientific evidence on the cost-effectiveness of PDNS care. Consequently, many hospitals lack the nursing capacity to offer PDNS care to all patients, which creates unequal access to care and possibly avoidable disability and costs.

Objective: The investigators aim to study the (cost-)effectiveness of specialized nursing care provided by a PDNS as compared to no PDNS care for people with PD in all disease stages. To gain more insight into the used interventions and their effects, a subgroup analysis will be performed based on disease duration (diagnosis made <5, 5-10, or >10 years ago).

Methods: The investigators will perform an 18-month, single-blind, randomized controlled clinical trial in eight community hospitals in the Netherlands. A total of 240 people with idiopathic PD that have not been treated by a PDNS over the past two years will be included, independent of disease severity or duration. In each hospital, 30 patients will randomly be allocated in a 1:1 ratio to either PDNS care according to the Dutch Guideline on PDNS care or no nursing intervention (continuing usual care). For the allocation of participants, a computer-generated list of random numbers will be used. The co-primary outcome measures are Quality of Life (QoL) and motor symptoms. Secondary outcomes include PD symptoms, mobility, non-motor symptoms, health-related quality of life, experienced quality of care, self-management, medication adherence, caregiver quality of life, coping skills and caregiver burden. Data will be collected after 12 months and 18 months. A healthcare utilization and productivity loss questionnaire will be completed every 3 months by both the patient and the caregiver.

Hypothesis: The investigators hypothesize that, by offering more patients access to PDNS care, QoL will increase with equal healthcare costs. Increasing direct medical costs (for nurse staffing) will be offset by a reduced number of consultations with the general practitioner and neurologist. If these outcomes are reached, wide implementation of PDNS care is needed.

DETAILED DESCRIPTION:
1. Background The Parkinson's Disease Nurse Specialist (PDNS) can fulfill a pivotal role in the multidisciplinary team of people with PD. The PDNS was introduced in 1989 in the United Kingdom to bridge the gap between medical management and the unique personal needs of patients. To obtain greater uniformity in care delivery by a PDNS and to facilitate the efficacy of nursing care in PD, the Dutch Guideline 'Nursing care in Parkinson's disease' was published in 2016. The main roles of the PDNS are clearly described in the Guideline, and include 1) providing information, education and instruction; 2) supporting the patient and caregiver in the promotion of self-management; 3) supporting psychosocial care questions; 4) prevention; 5) specialized diagnostic strategies and therapeutic nursing interventions; and 6) multidisciplinary collaboration.

   Based on expert opinion from healthcare professionals, the Dutch guideline advises that every person with PD could benefit from PDNS care, including those in early-stage disease where delivery of information, education about medication compliance and support in self-management are critical. So far, only three studies have evaluated PDNS care and they have found inconsistent results. Overall, they indicate that PDNS care may improve patient wellbeing, physical functioning and general health status and reduce anxiety and depression, but definite conclusions could not be drawn. Moreover, there is little evidence that shows that quality of life actually improves with PDNS care and to date, no studies have been performed that evaluated the cost-effectiveness of PDNS care.

   Currently, most hospitals in The Netherlands offer PDNS care, since it is advised in the Dutch Multidisciplinary Guideline. However many centers still lack the nursing capacity to offer PDNS care to all patients because the scientific evidence is inconclusive. This situation creates an undesirable inequality in access to care and presumably leads to avoidable disability and costs (e.g. from early admissions to nursing homes or crisis admissions to the hospital). Therefore, the investigators aim to study the cost-effectiveness of specialized nursing care provided by a PDNS as compared to no PDNS care for people with PD.
2. Study design The NICE-PD study is an 18-month, single-blind randomized controlled clinical trial that will be performed in eight community hospitals in the Netherlands. A total of 240 people with PD will be included (120 in each group) and equally distributed over the participating hospitals. The investigators have selected hospitals where, due to lack of sufficient PDNS staff, only a proportion of PD patients currently has access to PDNS care. This provides the investigators with a unique opportunity to identify patients who at present have no access to PDNS care, and to randomize them within hospitals (at the patient level) between PDNS care and no nursing intervention.

   Eligible patients will be allocated randomly to either PDNS care or usual care in a 1:1 ratio, using a computer-generated list of random numbers. To ascertain an equal representation of patients, the investigators will stratify for disease duration (according to pre-defined subgroups, i.e. disease duration <5 years, 5-10 years and >10 years). The PDNS intervention will be carried out according to the Dutch 'Guideline Nursing care in PD'. A blinded researcher will perform the clinical assessments at baseline (t0), after 12 months (t1) and after 18 months (t2). Patients and caregivers will also be asked to complete a set of questionnaires at t0, t1 and t2. Finally, every three months patients and their caregivers will complete an online questionnaire about healthcare utilization, costs and productivity loss.
3. Intervention

   The PDNS intervention will be performed according to the Dutch 'Guideline Nursing care in PD' published in 2015. The intervention is not standardized, but tailored to the patients' and caregivers' needs. This includes the following:
   * Assessment of individual care needs of people with PD and their caregivers. The PDNS performs a specific nursing assessment related to the medical, physical, psychological and social domains.
   * Development of a patient-centered treatment plan that supports the patient and caregiver in self-management. The PDNS composes a multidisciplinary plan, based on the results of the individual assessment, and as prioritized by the patient and caregiver (shared decision making). The treatment plan is developed according to the national self-management framework.
   * Specific nursing interventions. The intervention varies across disease stages and is tailored to the specific problems and needs of individual patients and their caregivers. The Guideline on PDNS care describes general- and specific nursing interventions. General interventions consist of providing information and education, disease management (e.g. considering advanced treatment options such as DBS) and monitoring (e.g. of caregiver burden). Specific nursing interventions are described for the following areas: mental functions, fatigue, sleep, urogenital functions, sexuality, medication adherence, orthostatic hypotension, caregiver burden, coping, mobility, self-management and dietary issues (table 2 provides examples of such interventions).
   * Collaboration with other healthcare professionals. The PDNS stimulates and supports multidisciplinary collaboration between healthcare professionals based on the individual patient-centered treatment plan. The PDNS also plays a pivotal role in the timely referral to other healthcare professionals.

   The PDNS will keep a pre-defined electronic study report according to a structured format for each PD patient, documenting the individual care needs, present symptoms, performed interventions and (changes in) the individual care plan. This report will be started at the initial assessment and updated at every follow-up contact with the patient, e.g. at the outpatient clinic, during a telephone consultation or at a home visit. This data will be purposefully collected for a possible process analysis at the end of the study.

   Patients will have regular contact with their PDNS about the progress and realization of the personal goals, both during face-to-face contacts and by telephone, and sometimes during additional home visits. The frequency and type of contact will be optimized for each patient depending on disease stage and individual patient needs. The Guideline on PDNS care advises that each patient has a minimum of one contact with the PDNS each year. Currently in the Netherlands, patients are seen on average twice a year by their PDNS, with an additional two interim telephone consultations per year.

   The control group will receive ongoing/ usual care which is otherwise comparable, but without a nursing intervention. This involves regular consultations with a neurologist in their own community hospital (typically 2-4 times per year, depending on patient preferences and health status). In addition, control patients will have no other restrictions considering any other medical treatments (e.g. by a psychologist or social worker). Importantly, many important elements of care (including in particular the treating neurologist) remain comparable between the two intervention arms because of the randomization at patient level within hospitals.
4. Clinical assessments At baseline, t1 and t2 all patients will visit their own hospital for the study assessments which are performed by a blinded researcher (PDQ-39, MDS-UPDRS, and TUG). Furthermore, the patients and their caregivers will complete additional home questionnaires. In addition, every three months, patients will receive a questionnaire at home regarding healthcare utilization, costs and productivity loss over the past three months. Caregivers will complete a cost questionnaire including healthcare utilization, costs and productivity loss specifically related to caregiver burden. Patients can choose if they want to fill out digital or paper questionnaires.
5. Data analysis The economic evaluation investigates, alongside the clinical trial, the value for money of full implementation of the PDNS into PD care from a societal and healthcare perspective. The investigators will take all relevant costs into account. The cost-effectiveness timeframe adheres to the clinical study protocol and evaluates cost-effectiveness up to 18 months after randomization. Cost will be measured using a healthcare utilization questionnaire (e.g. including medical consultations, hospital admissions, medication, travel costs, etc.) and a questionnaire measuring productivity loss while working of both patients and caregivers. Per item of healthcare consumption, standard cost-prices will be determined using the guideline for performing economic evaluations. If standardized prices are not available, full cost prices will be determined using activity based costing. Costs will be analyzed using a mixed model approach or a general linear model approach with a gamma distribution using a log link to account for possible skewness of the cost data.

   The investigators will use a PD-specific quality of life measure (PDQ-39) and a generic health-related quality of life scale (EQ5D) to evaluate the quality of the health status of patients. The potential difference in Quality-Adjusted Life Years (QALYs) measured with the EQ5D will be analyzed with a regression approach. The investigators will use a linear mixed model with repeated measurements to test for differences in quality of life (measured with the PDQ-39) between both groups. The same analysis will be used to measure differences between groups in the secondary outcome measures. The investigators will include study center as a random effect and fixed effects for group, time and the interaction between group and time. Each of the outcomes will be included as dependent variable. Statistical analyses will be performed based on the intention-to-treat principle.

   Besides the overall cost-effectiveness evaluation, the investigators will perform a pre-planned subgroup analysis based on disease duration (diagnosis made <5 years, 5-10 years or >10 years ago) to obtain more insight into the nursing interventions used in each disease stage and the effects of PDNS care in these different groups of patients. This subgroup analysis will be performed because, for example, for the more severely affected patients the nursing intervention is expected to become more intensive and possibly more effective, but also more expensive. When different patterns of this kind are found, this should be investigated further in future trials that are powered adequately to address such group differences.
6. Discussion The investigators hypothesize that offering PDNS care will lead to higher quality of life with equal healthcare costs. Increasing direct medical costs (for nurse staffing) are expected to be offset by a reduced number of (telephone) consultations with the general practitioner and neurologist. These short-term goals are the focus of the present NICE-PD proposal. In addition to the short-term effects, the investigators also expect long-term benefits, which are out of scope of the present project. Examples of potential long-term benefits include a reduction in the number of nursing home admissions and fewer emergency visits to the hospital, which would lead to a substantial cost reduction.

In conclusion, this study will generate new insights into the cost-effectiveness of specialized PD nursing interventions for people with PD. If positive results are found, a large shift in the organization of PD care is needed to warrant equal access to PDNS care for every person with PD.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of idiopathic PD;
* Sufficient knowledge of the Dutch language to fill out questionnaires;
* Age 18 years or older at the time of diagnosis;
* All disease stages, regardless of disease severity or disease duration;
* Not having received care from a PDNS in the past two years;
* A score of ≥ 18 on the Mini-Mental State Examination (MMSE13) and ≥ 12 on the Frontal Assessment Battery (FAB14).

Exclusion Criteria:

* A type of atypical parkinsonism caused by medication (e.g. neuroleptics), a metabolic disorder (e.g. Wilson's disease), encephalitis or a neurodegenerative disorder (e.g. multiple system atrophy, progressive supranuclear palsy, corticobasal syndrome).
* Residing in a nursing home or another type of residential care facility (because the PDNS is not operational there).
* Any other medical or psychiatric disorder that, in the opinion of the researcher, may compromise participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Disease-specific health-related quality of life: Parkinson's disease Questionnaire (PDQ-39) | Baseline, change from baseline quality of life at 12 months, change from baseline quality of life at 18 months
  Parkinson's disease Questionnaire (PDQ-39). Total score range: 0-100, including 8 subcategories. Subcategories are summed to compute the total score. A lower score means a better outcome.
Motor symptoms | Baseline, change from baseline motor symptoms at 12 months, change from baseline motor symptoms at 18 months
  Movement Disorders Society-sponsored revision of the Unified Parkinson's Disease Rating Scale part III (MDS-UPDRS part III). Total score range: 0-132. A lower score means a better outcome.

SECONDARY OUTCOMES:
Longitudinal Parkinson's disease symptoms | Baseline, change from baseline Parkinson's disease symptoms at 12 months, change from baseline Parkinson's disease symptoms at 18 months
  Movement Disorders Society-sponsored revision of the Unified Parkinson's Disease Rating Scale part I, II, IV (MDS-UPDRS part I, II, IV). Total score range: 0-260 (including the MDS-UPDRS part III), including 4 subcategories. Subcategories are summed to compute the total score. A lower score means a better outcome.
Mobility | Baseline, change from baseline TUG at 12 months, change from baseline TUG at 18 months
  Timed up and Go (TUG). A lower score means a better outcome.
Non-motor symptoms (anxiety and depression) | Baseline, 12 months, 18 months
  Hamilton Anxiety and Depression Scale (HADS). Total score range: 0-21, including 2 subcategories. Subcategories are summed to compute the total score. A lower score means a better outcome.
Non-motor symptoms | Baseline, change from baseline at 12 months, change from baseline at 18 months
  Scales for Outcomes in Parkinson's disease - Autonomic Questionnaire (SCOPA-AUT). Total score range: 0-69, including 6 subcategories. Subcategories are summed to compute the total score. A lower score means a better outcome.
Health-related quality of life: EuroQoL5D (EQ5D) | Baseline, change from baseline at 12 months, change from baseline at 18 months
  EuroQoL5D (EQ5D). Summary index with a maximum score of 1, including 5 dimensions. A higher score means a better outcome. In addition, there is a visual analogue scale (VAS) to indicate general health status with a total score range of 0-100. A higher score means a better outcome.
Experienced quality of and experience with provided healthcare: Consumer Quality Index (CQI) | Baseline, change from baseline at 12 months, change from baseline at 18 months
  Consumer Quality Index (CQI). There is no minimum or maximum score (the measure consists of a number of qualitative and experience questions). Therefore, higher values do not correlate with a better or worse outcome.
Self-management | Baseline, change from baseline at 12 months, change from baseline at 18 months
  Patient Activation Measure (PAM13). Total score range: 0-100, including a division in 4 activation levels. A higher score means a higher activation level (= the patient has made most of the necessary behavior changes to manage their disease).
Medication adherence | Baseline, change from baseline at 12 months, change from baseline at 18 months
  Morisky Medication Adherence Scale (MMAS). Total score range: 0-8. A higher score means a better outcome.
Health-related quality of life of the caregiver: EuroQoL5D (EQ5D) | Baseline, change from baseline at 12 months, change from baseline at 18 months
  EuroQoL5D (EQ5D). Summary index with a maximum score of 1, including 5 dimensions. A higher score means a better outcome. In addition, there is a visual analogue scale (VAS) to indicate general health status with a total score range of 0-100. A higher score means a better outcome.
Caregiver burden | Baseline, change from baseline at 12 months, change from baseline at 18 months
  Zarit Caregiver Burden Index (ZBI). Total score range: 0-88. A lower score means a better outcome.
Caregiver quality of life: CarerQol-7D | Baseline, change from baseline at 12 months, change from baseline at 18 months
  CarerQol-7D. Total score range: 0-14 (weighted sum score: 0-100). A higher score means a better outcome. In addition, there is a visual analogue scale (VAS) to indicate general well-being with a total score range of 0-10. A higher score means a better outcome.
Skills of proactive coping of the caregiver | Baseline, change from baseline at 12 months, change from baseline at 18 months
  Utrecht Proactive Coping Competence Scale (UPCC). Total score range: 21-84. A higher score means a better outcome.
Medical consumption of the patient | Baseline, change from baseline at 3 months, 6 months, 9 months, 12 months, 15 months and 18 months
  Medical Consumption Questionnaire (MCQ). There is no minimum or maximum score, this scale is a generic instrument for measuring medical costs.
Productivity loss of the patient | Baseline, change from baseline at 3 months, 6 months, 9 months, 12 months, 15 months and 18 months
  Productivity Cost Questionnaire (PCQ). There is no minimum or maximum score, this scale is a generic instrument to measure productivity losses related to the disease.
Medical consumption of the caregiver related to providing care to the patient | Baseline, change from baseline at 3 months, 6 months, 9 months, 12 months, 15 months and 18 months
  Adjusted version of the Medical Consumption Questionnaire (MCQ). There is no minimum or maximum score, this scale is a generic instrument for measuring medical costs.
Productivity loss of the caregiver related to providing care to the patient | Baseline, change from baseline at 3 months, 6 months, 9 months, 12 months, 15 months and 18 months
  Adjusted version of the Productivity Cost Questionnaire (PCQ). There is no minimum or maximum score, this scale is a generic instrument to measure productivity losses related to being a caregiver.
Nighttime sleep problems and daytime sleepiness | Baseline, change from baseline at 12 months, change from baseline at 18 months
  Scales for Outcomes in Parkinson's disease - Sleep Questionnaire (SCOPA-SLEEP). Total score range: 0-33, including 2 subcategories. Subcategories are summed to compute the total score. A lower score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Bastiaan R Bloem, MD, PhD, Principal Investigator — Department of Neurology, Radboudumc, Nijmegen, The Netherlands.
Locations (1):
- Radboud University Medical Center, Department of Neurology, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lennaerts H, Groot M, Rood B, Gilissen K, Tulp H, van Wensen E, Munneke M, van Laar T, Bloem BR. A Guideline for Parkinson's Disease Nurse Specialists, with Recommendations for Clinical Practice. J Parkinsons Dis. 2017;7(4):749-754. doi: 10.3233/JPD-171195. PMID 28800338
- [Background] Jahanshahi M, Brown RG, Whitehouse C, Quinn N, Marsden CD. Contact with a nurse practitioner: a short-term evaluation study in Parkinson's disease and dystonia. Behav Neurol. 1994;7(3):189-96. doi: 10.3233/BEN-1994-73-414. PMID 24487336
- [Background] Reynolds H, Wilson-Barnett J, Richardson G. Evaluation of the role of the Parkinson's disease nurse specialist. Int J Nurs Stud. 2000 Aug;37(4):337-49. doi: 10.1016/s0020-7489(00)00013-4. PMID 10760541
- [Background] Jarman B, Hurwitz B, Cook A, Bajekal M, Lee A. Effects of community based nurses specialising in Parkinson's disease on health outcome and costs: randomised controlled trial. BMJ. 2002 May 4;324(7345):1072-5. doi: 10.1136/bmj.324.7345.1072. PMID 11991913
- [Derived] Radder DLM, Lennaerts HH, Vermeulen H, van Asseldonk T, Delnooz CCS, Hagen RH, Munneke M, Bloem BR, de Vries NM. The cost-effectiveness of specialized nursing interventions for people with Parkinson's disease: the NICE-PD study protocol for a randomized controlled clinical trial. Trials. 2020 Jan 15;21(1):88. doi: 10.1186/s13063-019-3926-y. PMID 31941538
- See also: Dutch Multidisciplinary Guideline for Parkinson's disease — http://parkinsonnet.info/media/2733747/7994_multidisciplin_rl_parkinson_c_-_2011.pdf

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT03830190/Prot_SAP_000.pdf